CLINICAL TRIAL: NCT07363486
Title: Prospective Sequential Study of Dose-Escalating 225Ac-LNC1011 in the Treatment of Metastatic Castration-Resistant Prostate Cancer
Brief Title: Sequential Study of 225Ac-LNC1011 in the Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sequential Study-225Ac-LNC1011
Record Dates: First submitted 2025-12-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3.70 MBq (100 μCi) 225Ac-LNC1011 dose cohort (Experimental): Participant will receive 3.70 MBq (+/- 10%) 225Ac-LNC1011, once every 8-12 weeks for up to 4 cycles
  Interventions: Drug: 225Ac-LNC1011
- 5.55 MBq (150 μCi) 225Ac-LNC1011 dose cohort (Experimental): Participant will receive 5.55 MBq (+/- 10%) 225Ac-LNC1011, once every 8-12 weeks for up to 4 cycles
  Interventions: Drug: 225Ac-LNC1011
- 7.40 MBq (200 μCi) 225Ac-LNC1011 dose cohort (Experimental): Participant will receive 7.40 MBq (+/- 10%) 225Ac-LNC1011, once every 8-12 weeks for up to 4 cycles
  Interventions: Drug: 225Ac-LNC1011

INTERVENTIONS:
Drug: 225Ac-LNC1011 — administered intravenously once every 8-12 weeks (1 cycle) for up to 4 cycles

SUMMARY:
PSMA is an ideal target for the precise diagnosis and treatment of prostate cancer. LNC1011 is a novel albumin-binding PSMA-targeted compound. This study aims to investigate the safety and efficacy of different doses of 225Ac-labeled LNC1011 in the treatment of patients with PSMA-positive metastatic castration-resistant prostate cancer (mCRPC) and to explore the optimal therapeutic dose.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA)-targeted radioligand therapy has demonstrated considerable potential in the treatment of metastatic castration-resistant prostate cancer (mCRPC). By incorporating albumin-binding motifs into PSMA radioligands, the circulation time in the bloodstream can be prolonged, leading to significantly enhanced tumor uptake and therapeutic efficacy. LNC1011 employs dansylated Amino Acid as a novel, relatively weak yet high-performance albumin-binding moiety, achieving an optimal balance among increased tumor accumulation, improved safety, and refined diagnostic performance. This enables a unified theranostic approach within a single molecular framework.

Alpha-emitting radionuclides, represented by Ac-225, generate alpha particles during decay. Their linear energy transfer is nearly 100-fold higher than that of β-emitters such as Lu-177, resulting in significantly enhanced tumor cell kill. This has earned them the designation of "scalpel-like radiotherapy." Moreover, alpha particles have an extremely short range (only a few cell diameters), causing minimal damage to surrounding normal tissues and almost no notable side effects, thereby conferring an excellent safety profile.

In this clinical study, we will follow a "3+3" trial design to evaluate the safety and efficacy of different doses of 225Ac-LNC1011 in patients with mCRPC. The initial dose of 225Ac-LNC1011 is set at 3.70 MBq (100 μCi). Approximately three subjects will be enrolled at the current dose level. If no dose-limiting toxicity (DLT) is observed, the next cohort will receive an escalated dose of 5.55 MBq (150 μCi). If again no DLT occurs, the subsequent cohort will be escalated to 7.40 MBq (200 μCi), which is the planned maximum dose. It should be noted that if one DLT occurs at any dose level, three additional patients will be enrolled at the same dose. If only one DLT is observed among the total of six subjects, dose escalation may proceed. If two or more DLTs occur, dose de-escalation or trial termination will be initiated. Subjects in all dose cohorts will receive up to four treatment cycles at 8- to 12-week intervals. All participants will undergo safety follow-up during the trial and for 12 months after its completion.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic Castration-Resistant Prostate Cancer (mCRPC) mCRPC refers to prostate cancer that progresses despite serum testosterone at castrate levels (< 50 ng/dL or 1.7 nmol/L), meeting at least one of the following criteria:

   * PSA >1 ng/mL with two consecutive rises at least 1 week apart, each increase ≥50% above the nadir.
   * Radiographic progression: Either two or more new bone lesions on bone scan, or soft tissue lesion progression as per RECIST 1.1 criteria. Progression based on symptoms alone is insufficient for mCRPC diagnosis and requires further evaluation.
2. Failure of, Refusal of, Absence of, or Refractoriness to Standard Therapy, or Disease Progression, or No Available Standard Therapy per Current Guidelines:

   * Patients who have not received, refused, or progressed after receiving at least 1 but no more than 2 prior taxane-based therapies. The taxane regimen must have included exposure for at least 2 cycles. Patients who received only one taxane may be included if the investigator deems them unsuitable for a second taxane (e.g., due to frailty assessed by geriatric/comorbidity evaluation or intolerance).
   * Patients who have progressed after receiving at least one novel androgen axis drug [NAAD] (e.g., abiraterone, enzalutamide).
3. Ability to understand and voluntarily sign a written informed consent form (ICF), and willingness and ability to comply with trial procedures including examinations and follow-up.
4. Age 18-90 years (inclusive).
5. Expected survival > 6 months.
6. ECOG performance status ≤ 2.
7. Presence of high-uptake lesions confirmed by 68Ga-PSMA-11 PET/CT imaging (positive defined as lesion uptake >1.5 times the liver background).
8. At least one measurable lesion per RECIST 1.1 criteria OR at least one bone metastasis per PCWG3 criteria.
9. Adequate organ function (No blood products, growth factors, or albumin administered within 14 days prior to baseline lab tests):

   * Bone Marrow Function: Neutrophil count ≥ 1.5 × 10#/L, White blood cell count ≥ 3.0 × 10#/L, Platelet count ≥ 100 × 10#/L, Hemoglobin ≥ 10 g/dL (≥ 100 g/L).
   * Liver Function: Albumin ≥ 30 g/L, Total bilirubin ≤ 1.5 × ULN, ALT or AST ≤ 3.0 × ULN (without liver metastases) or ≤ 5.0 × ULN (with liver metastases).
   * Renal Function: Serum creatinine ≤ 1.5 × ULN.
   * Coagulation: INR ≤ 1.5; Activated partial thromboplastin time (APTT) ≤ 2 × ULN (for patients not on anticoagulation or on stable-dose anticoagulation).
10. Agreement to comply with prescribed radiation protection measures during the trial period.

Exclusion Criteria:

1. Inability to tolerate imaging procedures;
2. Patients who have received systemic anticancer therapy (e.g., chemotherapy, radiotherapy, immunotherapy; excluding endocrine therapy), investigational drugs, or device therapy within 4 weeks prior to dosing;
3. Patients who received radionuclide therapy (Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, Lutetium-177) within 6 months, or any External Beam Radiation Therapy (EBRT) within 2 months prior to the first dose;
4. Patients with unresolved Grade 4 myelosuppression from prior anticancer therapy within 2 weeks, or Grade 3 myelosuppression requiring >6 weeks for recovery;
5. Planned use of cytotoxic chemotherapy, antitumor immunotherapy, radioligand therapy, or similar agents during the study;
6. Use of blood products or albumin within 14 days before dosing to meet enrollment criteria;
7. Brain metastasis at screening, except:

   * Asymptomatic cases confined to supratentorial/cerebellar regions (no midbrain/pons/medulla/spinal cord involvement) without corticosteroid therapy and with lesions ≤1.5 cm;
   * Symptomatic cases with treated and radiologically stable lesions (>4 weeks);
8. Other malignancies within 5 years (excluding cured localized cancers like basal/squamous cell skin carcinoma);
9. Superscan on bone scintigraphy;
10. Symptomatic or impending spinal cord compression;
11. Prior EBRT involving extensive bone marrow (>25%);
12. Significant cardiac disease at screening, including:

    * QTcF >470 ms or long QT syndrome history;
    * Myocardial infarction, angina, or CABG within 6 months deemed ineligible by investigators;
13. Any condition that, per investigator judgment, may compromise safety, data interpretation, or indicate high risk;
14. Uncontrolled bladder outlet obstruction, urinary incontinence, claustrophobia, or radiophobia at screening;
15. Positive for HCV-Ab, HIV, or syphilis antibodies at screening;
16. HBsAg-positive patients with active HBV replication (confirmed by HBVDNA per investigator assessment);
17. Known allergy to proteins/peptides, excipients, or structurally related compounds;
18. History of drug/alcohol abuse within 1 year or chronic substance abuse;
19. Failure to use effective contraception during the trial and for 6 months post-last dose;
20. Severe active infection prior to the first administration.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events | From enrollment till 30 days safety follow-up, assessed up to 50 months (estimated final OS analysis)
  The distribution of adverse events (AE) will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Prostate-specific antigen 50 (PSA50) response | From date of randomization till 30 days safety fup, assessed up to 50 months (estimated final OS analysis)
  PSA50 response is defined as the proportion of patients who have a more/equal 50% decrease in PSA from baseline, it will be calculated at 12, 24 and 48 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of enrollment until date of progression or date of death from any cause, whichever come first, assessed up to 50 months (estimated final OS analysis)
  PSA-PFS is defined as the time from date of enrollment to the date of first documented progression by investigator assessment (radiographic progression, clinical progression, PSA progression) or death from any cause, whichever occurs first

OTHER OUTCOMES:
Overall Survival (OS) | From date of enrollment until date of death from any cause, assessed up to 50 months (estimated final OS analysis)
  OS is defined as time to death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Study Chair — Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China